CLINICAL TRIAL: NCT04960917
Title: Development and Implementation of eHealth Literacy Workshops in the Community
Brief Title: eHealth Literacy Workshops in the Community
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: eHL-HMO-CTIL
Record Dates: First submitted 2021-06-28; First posted 2021-07-14 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Health Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eHealth literacy workshop (Experimental): Community members from pre-existing municipality groups will participate in a workshop aimed to raise their ehealth literacy level.
  Interventions: Behavioral: Evaluation of ehealth literacy workshop

INTERVENTIONS:
Behavioral: Evaluation of ehealth literacy workshop — Intervention components will include a three session workshop, enabling participants to raise their knowledge of the different available health resources and how to find them, their ability to determine which health resource is reliable, their ability to use the health information online to make health decisions, their knowledge of the online services offered by HMOs/Ministry of Health, and their ability to navigate HMO and preform actions such as set an appointment, find a doctor, and find contact information

SUMMARY:
This study aims to implement and evaluate an eHeath literacy workshop that trains women to take advantage of the digital media available to them so that they can use it to their advantage- set appointments, search for doctors, critically read and understand health information, search for information about medications, diseases, health habits and more.

DETAILED DESCRIPTION:
This study aims to implement and evaluate an eHeath literacy workshop that trains women to take advantage of the digital media available to them so that they can use it to their advantage- set appointments, search for doctors, critically read and understand health information, search for information about medications, diseases, health habits and more. A three-session workshop (each session 1.5-2 hours) will take place via the web (for example -on zoom), or as a frontal workshop, (if MOH guidelines permitting due to COVID-19). The groups will have up to 20 participants, taking into account dropout rates of target population. Data will be collected at the first session, and at the last session. This program offers an interactive ehealth literacy workshop for men and women ages 45-75. The workshop, given by Pollin Center staff, will provide participants with the skills and tools to enable safe web surfing, search effectively for information, identify credible health information, as well as critically read and understand online information. It will also empower participants with the confidence and ability to use the information they access in achieving better personal health - allowing them to actively engage in their own care. Additionally, the workshop will review the basic services provided by HMO platforms, including the option to make appointments and search for other HMO services.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 45-76
* Must be able to read and write in Hebrew
* Must have access to the internet
* Must have basic computer skills (including web surfing, information searching, and basic website navigation skills).

Exclusion Criteria:

- Women and men who don't meet the above criteria.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in level of ehealth literacy | At baseline and immediately after the intervention (workshop)
  Level of eHealth literacy will be assessed by using the validated eHealth Literacy Scale, "eHEALS" (Norman and Skinner, 2006), a self report 8-item measure of eHealth literacy (score range: 8-40, higher score means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD, MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Tennant B, Stellefson M, Dodd V, Chaney B, Chaney D, Paige S, Alber J. eHealth literacy and Web 2.0 health information seeking behaviors among baby boomers and older adults. J Med Internet Res. 2015 Mar 17;17(3):e70. doi: 10.2196/jmir.3992. PMID 25783036
- [Background] Xie B. Effects of an eHealth literacy intervention for older adults. J Med Internet Res. 2011 Nov 3;13(4):e90. doi: 10.2196/jmir.1880. PMID 22052161
- [Background] Mitsutake S, Shibata A, Ishii K, Oka K. Associations of eHealth Literacy With Health Behavior Among Adult Internet Users. J Med Internet Res. 2016 Jul 18;18(7):e192. doi: 10.2196/jmir.5413. PMID 27432783
- [Background] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046